CLINICAL TRIAL: NCT01911052
Title: The Impact of Telephone and Short Message System Based Education on Bowel Preparation for Colonoscopy in Health Screened Population
Brief Title: The Impact of Telephone and Short Message System Based Education on Bowel Preparation for Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Kim Eun Soo, Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-05-050-002
Record Dates: First submitted 2013-07-22; First posted 2013-07-30 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Bowel Preparation
Keywords: Bowel preparation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention (Experimental): The investigational, or experimental arm, will receive standard written instructions on preparing for a colonoscopy plus intervention such as telephone based re-education by one investigator on the day before colonoscopy.
  Interventions: Other: Telephone based re-education
- Standard preparation instructions (No Intervention): The control arm will receive written instruction on preparing for a colonoscopy per standard of care at Keimyung University Dongsan Medical Center
- Interventional (Experimental): The investigational, or experimental arm, will receive standard written instructions on preparing for a colonoscopy plus intervention such as short message system based re-education by one investigator on the day before colonoscopy.
  Interventions: Other: Short message system based re-education

INTERVENTIONS:
Other: Telephone based re-education — The investigational, or experimental arm, will receive standard written instructions on preparing for a colonoscopy plus intervention such as telephone based re-education by one investigator on the day before colonoscopy.
  Arms: Intervention
Other: Short message system based re-education — The investigational, or experimental arm, will receive standard written instructions on preparing for a colonoscopy plus intervention such as short message system based re-education by one investigator on the day before colonoscopy.
  Arms: Interventional

SUMMARY:
Inadequate bowel preparation results in decreased rates of cecal intubation, increased rates of missing important lesions, increased patient discomfort, higher risk of complications, prolonged procedure time and increased health-care cost. Recent study reported that Telephone-based re-education (TRE) on the day before colonoscopy significantly improved the quality of bowel preparation and polyp detection rate. However, there is no study to compare the effect of telephone with short message system (SMS) based re-education on the quality of bowel preparation in health screened population. Our goal is to improve the quality of bowel preparation with telephone or SMS based re-education for outpatients undergoing screening colonoscopies. The investigators hypothesise that efforts to improve education and maximise patient compliance during the preparatory period will enhance the efficacy of bowel preparation.

ELIGIBILITY:
Inclusion Criteria:

* All health screened populations
* age >18
* scheduled for an elective screening colonoscopy

Exclusion Criteria:

* inpatients
* pregnancy
* breast feeding
* prior history of surgical large bowel resection
* patients allergic to PEG-ELS based laxatives

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Quality of bowel preparation | day 1
  The primary outcomes will be the endoscopist's assessment of the quality of preparation using Boston and Ottawa bowel preparation scare

SECONDARY OUTCOMES:
polyp detection rate | day 1
  The number of polyp prescribed by endoscopist.

OTHER OUTCOMES:
Patient compliance | baseline
  Patient compliance with preparation instructions self-reported in a pre-procedure questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eun Soo Kim, Professor, Principal Investigator — Keimyung University School of Medicine
Locations (1):
- Eun Soo Kim, Daegu, South Korea

REFERENCES:
- [Background] Liu X, Luo H, Zhang L, Leung FW, Liu Z, Wang X, Huang R, Hui N, Wu K, Fan D, Pan Y, Guo X. Telephone-based re-education on the day before colonoscopy improves the quality of bowel preparation and the polyp detection rate: a prospective, colonoscopist-blinded, randomised, controlled study. Gut. 2014 Jan;63(1):125-30. doi: 10.1136/gutjnl-2012-304292. Epub 2013 Mar 16. PMID 23503044
- [Derived] Lee YJ, Kim ES, Choi JH, Lee KI, Park KS, Cho KB, Jang BK, Chung WJ, Hwang JS. Impact of reinforced education by telephone and short message service on the quality of bowel preparation: a randomized controlled study. Endoscopy. 2015 Nov;47(11):1018-27. doi: 10.1055/s-0034-1392406. Epub 2015 Jul 16. PMID 26182387